CLINICAL TRIAL: NCT07080580
Title: Effects of Vibration-Assisted Core Stabilization Exercises on Menstrual Symptoms, Pain, and Quality of Life in Women With Primary Dysmenorrhea: A Randomized Controlled Trial
Brief Title: Vibration-Assisted Core Exercises for Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ebru Aloğlu Çiftçi (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Ebru Aloğlu Çiftçi, Lecturer, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EAloglu02
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Dysmenorrhea Primary
Keywords: Vibration; dysmenorrhea primary; core exercise; whole body vibration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole Body Vibration (Experimental): The vibration group performed core exercises with vibration at 8 mm amplitude and 14 Hz frequency, 3 days a week for 8 weeks (24 sessions). Each session lasted 45-60 minutes, including a 10-minute warm-up (walking) and a 5-minute cool-down (stretching). Vibration time started at 15 minutes and increased to 30 minutes. Eight core exercises (bridge exercise, plank, cat-camel exercise, crunches, side-bends, heel drops, squats, half push-ups) were applied, with repetitions increased every 2 weeks: 8 reps in weeks 1-2, 10 reps in weeks 3-4, 12 reps in weeks 5-6, and 15 reps in weeks 7-8. A 30-second rest was given between exercises.
  Interventions: Behavioral: Core exercises performed simultaneously on a whole body vibration platform
- Control Group (No Intervention): No intervention was applied to the control group.

INTERVENTIONS:
Behavioral: Core exercises performed simultaneously on a whole body vibration platform — It's a method where individuals stand on a vibration-generating platform and the vibration is transmitted from the soles of their feet to the entire body. Its use in combination with exercise has become popular in recent years due to the hypergravity it creates, aiming to increase muscle strength and reduce pain.
  There is no standardized protocol for the frequency, amplitude, and frequency of vibration application. However, it is known that when applied at frequencies between 10-30 Hz, it has no negative side effects and is beneficial in managing pain. In our study, core exercises will be performed on a vibration platform at a frequency of 14 Hz with an amplitude of 8 mm.
  Arms: Whole Body Vibration

SUMMARY:
This study aims to evaluate the effects of core stabilization exercises performed on a vibration platform in young women with primary dysmenorrhea. The exercises are designed to help reduce menstrual symptoms and pain, and to improve attitudes toward menstruation, functional and emotional well-being, and quality of life. A total of 24 women participated in the study. Participants were assigned either to a group receiving vibration-assisted core exercises or to a control group receiving no intervention. The intervention lasted 8 weeks, with sessions held three times per week.

DETAILED DESCRIPTION:
Primary dysmenorrhea (PD) is a common gynecological condition characterized by uterine-origin lower abdominal pain during or before menstruation in the absence of any pelvic pathology. This randomized controlled trial aims to investigate the effects of a core exercise (CE) program performed on a vibration-supported platform on pain intensity, menstrual attitudes, quality of life, and functional and emotional status in women with PD. A total of 24 women aged 18 to 35 years participated in the study. Participants were randomly assigned to either an intervention group (n=12) or a control group (n=12). The intervention group performed vibration-assisted CE on a portable platform three times per week for eight weeks. The control group received no intervention. All participants were evaluated within the first 48 hours of the menstrual cycle, with follow-up assessments at weeks 4, and a final evaluation at the end of week 8.

ELIGIBILITY:
Inclusion Criteria:

1. Being in the 18-28 age group.
2. Being diagnosed with primary dysmenorrhea on an ultrasound examination.
3. Having a Body Mass Index (BMI) between 19-24.9.
4. Describing pain intensity as 5 or higher on the VAS pain scale.
5. Having regular menstrual cycles (every 21-35 days and no intermenstrual bleeding) for the past 6 months.
6. Being willing to participate in the study.
7. Being cooperative and oriented.
8. Not having had any fractures, dislocations, or joint injuries in the past 6 months.
9. Not having had any surgery in the past 6 months.

Exclusion Criteria:

1. Having a systemic or chronic disease,
2. Being a professional athlete,
3. Having secondary dysmenorrhea,
4. Using oral contraceptives,
5. Being pregnant,
6. Having an orthopedic, neurological, rheumatological, or cardiovascular problem that prevents exercise,
7. Having any balance problems (vertigo, etc.) that prevent exercise.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Functional and Emotional Status Assessment (Functional and Emotional Dysmenorrhea Scale) | First 48 hours of the menstrual cycle (pre-intervention), week 4 (post-intervention), week 8 (post-intervention)
  The Functional and Emotional Dysmenorrhea Scale was used to assess participants' dysmenorrhea experiences functionally and emotionally. The scale is a Likert-type scale consisting of 14 items and two subscales. Each item can be scored from 1 to 5. Scoring criteria are: 1. Not at all like my situation, 2. Not at all like my situation, 3. Both similar and not like my situation, 4. Similar to my situation, 5. Very similar to my situation. As the total score on the scale increases, the extent to which individuals are functionally and emotionally affected by dysmenorrhea also increases.
Menstruation Symptoms (Menstruation Symptom Scale) | First 48 hours of the menstrual cycle (pre-intervention), week 4 (post-intervention), week 8 (post-intervention)
  In our study, the Menstrual Symptom Scale, a useful tool for assessing menstrual symptoms in Turkish women and found to have adequate validity and reliability, was used to assess participants' symptoms. The scale consists of 22 items developed to assess dysmenorrhea and its symptoms. Each item can be scored from 1 to 5. Scoring criteria range from 1 (never) to 5 (always). It consists of three subscales: items 1-13 address negative effects/somatic complaints, items 14-19 address menstrual pain symptoms, and items 20-22 address coping strategies. The subscale score is calculated by calculating the total mean score of the items in the subscales. A higher mean score for a subscale indicates an increase in the severity of menstrual symptoms related to that subscale. The mean score calculated from the scale is directly proportional to the severity of menstrual symptoms.
Menstruation Attitudes (Menstruation Attitude Questionnaire) | First 48 hours of the menstrual cycle (pre-intervention), week 4 (post-intervention), week 8 (post-intervention)
  In our study, we used the Menstruation Attitude Questionnaire to measure attitudes toward menstruation in individuals with dysmenorrhea and varying socio-demographic characteristics. The scale is a Likert-type scale consisting of 33 items and 5 subscales. Each item is scored from 1 to 5. Scoring criteria range from 1 (Strongly disagree) to 5 (Strongly agree). The subscales and number of items are as follows: 1. Menstruation as a debilitating phenomenon (12 items); 2. Menstruation as a disturbing phenomenon (6 items); 3. Menstruation as a natural phenomenon (5 items); 4. Precognition/Anticipation of menstruation (5 items); and 5. Denial of the effects of menstruation (7 items). A high mean score on the Menstruation Attitude Questionnaire is directly proportional to the positive attitude toward menstruation.

SECONDARY OUTCOMES:
Pain Intensity (Visual Analog Scale) | First 48 hours of the menstrual cycle (pre-intervention), week 4 (post-intervention), week 8 (post-intervention)
  VAS is a frequently used assessment method for converting the intensity of pain, which cannot be measured numerically, into numerical data. Pain intensity is assessed on a scale from 0 to 10, with 0 indicating no pain and 10 indicating unbearable pain.
Quality of Life Assessment (Short Form-36 Scale) | First 48 hours of the menstrual cycle (pre-intervention), week 4 (post-intervention), week 8 (post-intervention)
  The SF-36 is a self-assessment tool consisting of eight subscales and 36 questions. This tool is grouped to assess participants' physical functioning (10 items), physical limitations (4 items), emotional limitations (3 items), pain limitations (2 items), vitality (4 items), social functioning (2 items), mental health (5 items), and general health (5 items). Each subscale can be scored from 0 to 100. In this scoring system, 0 represents the lowest quality of life, and 100 represents the best.
Trunk endurance assessment (Sorenson Test) | First 48 hours of the menstrual cycle (pre-intervention), week 4 (post-intervention), week 8 (post-intervention)
  In the Sorenson Test, participants were positioned prone, their pelvises positioned at the edge of the table, and their ankles were stabilized. The upper extremities were positioned next to the torso. The time the participant could maintain the horizontal position was measured with a stopwatch. The test was terminated if the position could not be maintained.
Trunk endurance assessment (Sit-up testi) | First 48 hours of the menstrual cycle (pre-intervention), week 4 (post-intervention), week 8 (post-intervention)
  In the sit-up test, the maximum number of correct repetitions that the subjects perform within a 30-second time period is recorded.
Trunk endurance assessment (Lateral Bridge Test-Right and Left) | First 48 hours of the menstrual cycle (pre-intervention), week 4 (post-intervention), week 8 (post-intervention)
  The Side Bridge Test was performed to assess the endurance of the spinal stabilizer muscles. Participants were positioned in a side-lying position. They were asked to lift their hips until the pelvis and trunk were horizontal. The time the position was maintained was measured with a stopwatch, and the assessment was performed on both sides.

CONTACTS AND LOCATIONS:
Overall Officials: EBRU ALOĞLU ÇİFTÇİ, Lecturer, Principal Investigator — Okan University
Locations (1):
- Istanbul Okan University, Istanbul, Tuzla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study will share de-identified, summary-level outcome data, including group-level means, standard deviations, effect sizes, and p-values derived from statistical analyses.
Supporting Information: Study Protocol, SAP
Time Frame: Summary-level data and supporting documents (e.g., study protocol and statistical analysis plan) will be available within 12 months following the final publication of study results.
Access Criteria: The study's outcome results, including group-level means, standard deviations, p-values, and effect sizes, as well as supporting materials such as the study protocol and statistical analysis plan, will be made available to qualified academic researchers upon reasonable request.

REFERENCES:
- [Background] Lefebvre G, Pinsonneault O, Antao V, Black A, Burnett M, Feldman K, Lea R, Robert M; SOGC. Primary dysmenorrhea consensus guideline. J Obstet Gynaecol Can. 2005 Dec;27(12):1117-46. doi: 10.1016/s1701-2163(16)30395-4. English, French. PMID 16524531
- [Background] Hoseini, M., Gharahtapeh, S. R., Jahazi, A. 2015 "Effect Of Vibration And Heat Combination On Primary Dysmenorrhea" Bali Medical Journal, 4(1), 12-16.